CLINICAL TRIAL: NCT00662142
Title: Effect of 8-Week Dietary DHA Supplementation on Cerebral Blood Flow and Metabolic Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05-12-13-03 (MARTEK)
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Healthy; Attention
Keywords: DHA; fMRI
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (1):
- 1 (Experimental): DHA 400 mg/day (200mg twice daily), vs DHA 1200 mg/day (400 mg three times daily), vs placebo; 1:1:1 ratio
  Interventions: Dietary Supplement: docosahexaenoic acid

INTERVENTIONS:
Dietary Supplement: docosahexaenoic acid — DHA 400 mg/day (200mg twice daily), vs DHA 1200 mg/day (400 mg three times daily), vs placebo; 1:1:1 ratio
  Other Names: DHA

SUMMARY:
The goal of this study is to determine if 8-week dietary treatment with the omega-3 fatty acid docosahexaenoic acid (DHA) improves attention performance and associated cortical activity and metabolism in 8 - 10 year old males that were not breast-fed during infancy.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects between the ages of 8 - 10 years.
2. Not breast-fed during infancy
3. Right hand dominant
4. Attending school at appropriate grade level
5. Normal body-mass index (BMI)
6. Ability and willingness to provide assent and informed, written consent from at least one biological parent.
7. Present with biological parent
8. No current general medical or psychiatric illness.
9. Medication free.
10. Normal intelligence as assessed by the Kaufman Brief Intelligence Test.
11. Willingness to maintain current dietary habits.

Exclusion Criteria:

1. Inability or unwillingness to provide consent.
2. Antecedent or concurrent serious medical illness.
3. A lifetime history of any significant axis I psychiatric disorder ( i.e. bipolar disorder, schizophrenia)
4. Patients who have received any psychoactive medications, current and lifetime.
5. Clinically unstable medical disease, including cardiovascular, hepatic insufficiency, severe renal impairment, gastrointestinal, pulmonary, metabolic, endocrine, obesity or other systemic disease.
6. History of seizures, excluding febrile seizures in childhood.
7. Patients requiring treatment with any drug which might obscure the action of study the study treatment.
8. Less than normal intelligence.
9. Pacemaker
10. Cerebral aneurysm clip
11. Cochlear implant
12. Metal fragments lodged within the eye
13. Claustrophobia
14. Necessity of sedation (no sedation will be given).
15. History of loss of consciousness > 10 minutes in duration
16. Adopted

Ages: 8 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
performance on sustained attention task (CPT-IP) | 8 weeks

SECONDARY OUTCOMES:
fMRI activation of prefrontal and frontal cortical regions during performance of an attention task (CPT-IP) | 8 weeks
NAA concentrations | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert McNamara, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] McNamara RK, Able J, Jandacek R, Rider T, Tso P, Eliassen JC, Alfieri D, Weber W, Jarvis K, DelBello MP, Strakowski SM, Adler CM. Docosahexaenoic acid supplementation increases prefrontal cortex activation during sustained attention in healthy boys: a placebo-controlled, dose-ranging, functional magnetic resonance imaging study. Am J Clin Nutr. 2010 Apr;91(4):1060-7. doi: 10.3945/ajcn.2009.28549. Epub 2010 Feb 3. PMID 20130094